CLINICAL TRIAL: NCT06918366
Title: A Randomized, Double-blind, Placebo-controlled Phase Ia Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of XQ-001 for Inhalation in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Inhaled XQ-001 in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brilliant Inspiration Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: XQ-2023CT-001-01
Record Dates: First submitted 2025-04-08; First posted 2025-04-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part A - single rising dose 1 (Other): inhalation
  Interventions: Drug: Part A - single rising dose 1
- Part A - single rising dose 2 (Other): inhalation
  Interventions: Drug: Part A - single rising dose 2
- Part A - single rising dose 3 (Other): inhalation
  Interventions: Drug: Part A - single rising dose 3
- Part A - single rising dose 4 (Other): inhalation
  Interventions: Drug: Part A - single rising dose 4
- Part A - single rising dose 5 (Other): inhalation
  Interventions: Drug: Part A - single rising dose 5
- Part A - single rising dose 6 (Other): inhalation
  Interventions: Drug: Part A - single rising dose 6
- Part B - multiple rising dose 1 (Other): inhalation
  Interventions: Drug: Part B - mutiple rising dose 1
- Part B - multiple rising dose 2 (Other): inhalation
  Interventions: Drug: Part B - mutiple rising dose 2

INTERVENTIONS:
Drug: Part A - single rising dose 1 — Inhaled XQ-001
  Other Names: Single dose 1
  Arms: Part A - single rising dose 1
Drug: Part A - single rising dose 2 — Inhaled XQ-001 or Placebo
  Other Names: Single dose 2
  Arms: Part A - single rising dose 2
Drug: Part A - single rising dose 3 — Inhaled XQ-001 or Placebo
  Other Names: Single dose 3
  Arms: Part A - single rising dose 3
Drug: Part A - single rising dose 4 — Inhaled XQ-001 or Placebo
  Other Names: Single dose 4
  Arms: Part A - single rising dose 4
Drug: Part A - single rising dose 5 — Inhaled XQ-001 or Placebo
  Other Names: Single dose 5
  Arms: Part A - single rising dose 5
Drug: Part A - single rising dose 6 — Inhaled XQ-001 or Placebo
  Other Names: Single dose 6
  Arms: Part A - single rising dose 6
Drug: Part B - mutiple rising dose 1 — Inhaled XQ-001 or Placebo
  Other Names: Mutiple dose 1
  Arms: Part B - multiple rising dose 1
Drug: Part B - mutiple rising dose 2 — Inhaled XQ-001 or Placebo
  Other Names: Mutiple dose 2
  Arms: Part B - multiple rising dose 2

SUMMARY:
The primary study objective is to evaluate the safety and tolerability of XQ-001 for inhalation after single and multiple nebulized inhalation administration in healthy Chinese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy adult male or female subjects aged 18-45 years old (including the boundary value, based on the time of signing the informed consent form) at the time of screening;
* 2) Body mass index (BMI: weight [kg]/height [m]2) is between 18.0 and 28.0 kg/m2 (inclusive), male subjects weigh ≥50 kg, and female subjects weigh ≥45 kg;
* 3) Normal lung function during the screening period, i.e., FEV1 ≥ 80% predicted and FEV1/FVC > 92% predicted;
* 4) During the screening period, the subjects' vital signs, physical examinations, laboratory tests, 12-lead electrocardiogram (ECG) and chest X-ray showed no abnormalities or abnormalities without clinical significance;
* 5) Qualified subjects of fertile potential must agree to use a medically approved contraceptive measure (such as intrauterine contraceptive device, contraceptive pills or condoms) during the trial and within 6 months after the trial. Specific contraceptive measures are shown in Appendix 1; and have no plans to donate sperm/eggs during the trial and within 6 months after the trial;
* 6) Subjects fully understand the purpose, nature, methods and possible adverse reactions of the trial, voluntarily participate and sign a written informed consent form, and can complete the study in accordance with the requirements of the protocol.

Exclusion Criteria:

* 1) Known severe allergic, non-allergic drug reaction, or multiple drug allergies, or known hypersensitivity reaction to the investigational product (active drug substance or drug product excipients);
* 2) The presence of symptoms or related medical history of any major disease, including but not limited to heart, liver, kidney disease or other acute or chronic gastrointestinal diseases, respiratory diseases, bone and joint diseases, as well as blood, endocrine, neurological, mental and other systemic diseases, or any other disease or physiological condition that may interfere with the results of the trial; any surgical condition or condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or any surgical condition or condition that may pose a hazard to the subjects participating in the trial; such as history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or difficulty urinating, peptic tract ulcer, history of gastrointestinal bleeding, etc;
* 3) Those who have been diagnosed with or are currently suffering from bronchial asthma, airway hyperresponsiveness, or have history of suspected asthma attacks;
* 4) Current chronic liver disease or a known history of liver or biliary abnormalities that the investigator determines may affect the trial results; liver function test results at screening are outside the normal range of the research center and are determined by the investigator to be abnormal and clinically significant (two replicate assessments are allowed at the investigator's discretion);
* 5) Current arrhythmia diseases (symptomatic or asymptomatic) or a history of arrhythmia determined by the investigator to be abnormal and clinically significant;
* 6) Clinically significant ECG abnormalities, including but not limited to second or third degree atrioventricular block, QRS complex prolongation of more than 120 msec, or QTc interval prolongation (QTcF>450 msec for male subjects and QTcF>470 msec for female subjects, see Appendix 2 for the formula);
* 7) Heart rate <50 or >100 beats/minute at screening, and determined by the investigator to be abnormal and clinically significant;
* 8) Severe infection occurred within 30 days before the first administration, including cellulitis, infectious pneumonia, sepsis, etc. For subjects with mild infection (such as mild upper respiratory tract infection), the investigator can determine whether they are suitable for inclusion;
* 9) Received live vaccination within 30 days before the first dose;
* 10) Suffered from a major clinically significant disease or underwent major surgery within 3 months before the first dose (except for outpatient minor surgeries), or expected to need major surgery during the trial;
* 11) Those with a known or suspected history of drug abuse within 2 years before screening, or drug abuse within 3 months before screening, or positive drug abuse screening during the screening period and baseline period;
* 12) Those who have used clinical trial drugs within 3 months before the first dose, or plan to participate in other interventional clinical trials during this study;
* 13) Those who have used any prescription drugs (including drugs that induce and inhibit liver drug enzymes), over-the-counter drugs, Chinese herbal medicines, and health products within 14 days before the first dose (or within 7 half-lives, whichever is the longest);
* 14) Those who donated blood or lost blood ≥400 mL within 3 months before screening; or donated blood or lost blood ≥200 mL within 1 month before screening; or planned to donate blood during the study;
* 15) Those who used food or beverages that may affect liver metabolism (such as star fruit, pomelo, grapefruit, etc.) within 7 days before the first dose;
* 16) Those who habitually use nicotine products or smoke (more than 5 cigarettes per day) within 3 months before screening, or those who do not agree to refrain from smoking or using nicotine products during the trial;
* 17) Drink more than 14 units of alcohol per week within 6 months before screening (1 unit of alcohol = 360 mL of beer or 45 mL of 40% alcohol by volume liquor or 150 mL of wine); or those who have a positive alcohol breath test during the baseline period; or those who do not agree to refrain from taking any alcoholic products during the trial;
* 18) Those who are unwilling to refrain from caffeinated beverages from 24 hours before the first dose until the end of this study;
* 19) Positive human immunodeficiency virus (HIV) antibody, or positive hepatitis B surface antigen, or positive hepatitis C antibody, or positive syphilis spirochete antibody;
* 20) Malignant tumor within 5 years before screening (excluding resected and cured carcinoma in situ, such as non-malignant melanoma skin cancer, etc.);
* 21) Pregnant or lactating women, or those with a positive pregnancy test during the screening period or hospitalization examination;
* 22) The investigator believes that it is not appropriate to participate in this study for scientific reasons, compliance reasons, or subject safety reasons;
* 23) Those who have previously used XQ-001 for inhalation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Number (%) of participants experiencing adverse events (AE) and serious adverse events (SAE) | Up to 9 days
Number (%) of participants with clinically relevant changes in 12-lead ECGs, vital signs, clinical laboratory parameters, physical examinations, or pulmonary function test | Up to 9 days

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 24 hours after first and last dose
Time of maximum observed concentration (Tmax) | Up to 24 hours after first and last dose
Area under the plasma concentration-time curve (AUC) from time 0 to time t, where t is the last time point at which the concentration is above the lower limit of quantification (AUC0-t) | Up to 24 hours after first and last dose

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chendu, China